CLINICAL TRIAL: NCT05496686
Title: First in Human Phase I Study of 225Actinium-MTI-201 (225Ac-MTI-201) in Metastatic Uveal Melanoma
Brief Title: Targeted Alpha Particle Radiotherapy for Metastatic Uveal Melanoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Modulation Therapeutics, Inc. (Industry)
Collaborators: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC 19868; MTI201-IA (Other: Modulation Therapeutics, Inc)
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Uveal Melanoma; Metastatic
Keywords: Uveal Neoplasms; Melanoma of the Uvea; Melanocortin 1 Receptor; MC1R; Peptide Receptor Radiotherapeutic; PRRT; Actinium-225-PRRT
MeSH Terms: conditions — Uveal Melanoma; Neoplasm Metastasis; Uveal Neoplasms

STUDY DESIGN:
Intervention Model Description: The continual reassessment method (CRM) will be used for this study. The dose escalation plan is for a doubling of the dose for doses 2 through 6, a 1.67-fold increase for doses 7 and 8, and a 1.33-fold increase for doses 9-12. This plan corresponds roughly to the modified Fibonacci dose escalation plan given by Penel and Kramar.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- 225Ac-MTI-201 4.7 microCi (Experimental): Cohort 1: Participants were administered a single dose of 4.7 microCi of 225Ac-MTI-201 via intravenous catheter, with up to 3 years of follow-up.
  Interventions: Drug: 4.7 microCi 225Ac-MTI-201
- 225Ac-MTI-201 9.5 microCi (Experimental): Cohort 2: Participants were administered a single dose of 9.5 microCi of 225Ac-MTI-201 via intravenous catheter, with up to 3 years of follow-up.
  Interventions: Drug: 9.5 microCi of 225Ac-MTI-201
- 225Ac-MTI-201 19 microCi (Experimental): Cohort 3: Participants were administered a single dose of 19 microCi of 225Ac-MTI-201 via intravenous catheter, with up to 3 years of follow-up.
  Interventions: Drug: 19 microCi of 225Ac-MTI-201
- 225Ac-MTI-201 38 microCi (Experimental): Cohort 4: Participants were administered a single dose of 38 microCi of 225Ac-MTI-201 via intravenous catheter, with up to 3 years of follow-up.
  Interventions: Drug: 38 microCi of 225Ac-MTI-201
- 225Ac-MTI-201 76 microCi (Experimental): Cohort 5: Participants were administered a single dose of 76 microCi of 225Ac-MTI-201 via intravenous catheter, with up to 3 years of follow-up.
  Interventions: Drug: 76 microCi of 225Ac-MTI-201
- 225Ac-MTI-201 152 microCi (Experimental): Cohort 6: Participants were administered a single dose of 152 microCi of 225Ac-MTI-201 via intravenous catheter, with up to 3 years of follow-up.
  Interventions: Drug: 152 microCi of 225Ac-MTI-201
- 225Ac-MTI-201 254 microCi (Experimental): Cohort 7: Participants were administered a single dose of 254 microCi of 225Ac-MTI-201 via intravenous catheter, with up to 3 years of follow-up.
  Interventions: Drug: 254 microCi of 225Ac-MTI-201
- 225Ac-MTI-201 424 microCi (Experimental): Cohort 8: Participants were administered a single dose of 424 microCi of 225Ac-MTI-201 via intravenous catheter, with up to 3 years of follow-up.
  Interventions: Drug: 424 microCi of 225Ac-MTI-201
- 225Ac-MTI-201 564 microCi (Experimental): Cohort 9: Participants were administered a single dose of 564 microCi of 225Ac-MTI-201 via intravenous catheter, with up to 3 years of follow-up.
  Interventions: Drug: 564 microCi of 225Ac-MTI-201
- 225Ac-MTI-201 750 microCi (Experimental): Cohort 10: Participants were administered a single dose of 750 microCi of 225Ac-MTI-201 via intravenous catheter, with up to 3 years of follow-up.
  Interventions: Drug: 750 microCi of 225Ac-MTI-201
- 225Ac-MTI-201 998 microCi (Experimental): Cohort 11: Participants were administered a single dose of 998 microCi of 225Ac-MTI-201 via intravenous catheter, with up to 3 years of follow-up.
  Interventions: Drug: 998 microCi of 225Ac-MTI-201
- 225Ac-MTI-201 1327 microCi (Experimental): Cohort 12: Participants were administered a single dose of 1327 microCi of 225Ac-MTI-201 via intravenous catheter, with up to 3 years of follow-up.
  Interventions: Drug: 1327 microCi of 225Ac-MTI-201

INTERVENTIONS:
Drug: 4.7 microCi 225Ac-MTI-201 — 4.7 microCi intravenous solution
  Other Names: 4.7 microCi 225Actinium-MTI-201
  Arms: 225Ac-MTI-201 4.7 microCi
Drug: 9.5 microCi of 225Ac-MTI-201 — 9.5 microCi intravenous solution
  Other Names: 9.5 microCi 225Actinium-MTI-201
  Arms: 225Ac-MTI-201 9.5 microCi
Drug: 19 microCi of 225Ac-MTI-201 — 19 microCi intravenous solution
  Other Names: 19 microCi 225Actinium-MTI-201
  Arms: 225Ac-MTI-201 19 microCi
Drug: 38 microCi of 225Ac-MTI-201 — 38 microCi intravenous solution
  Other Names: 38 microCi 225Actinium-MTI-201
  Arms: 225Ac-MTI-201 38 microCi
Drug: 76 microCi of 225Ac-MTI-201 — 76 microCi intravenous solution
  Other Names: 76 microCi 225Actinium-MTI-201
  Arms: 225Ac-MTI-201 76 microCi
Drug: 152 microCi of 225Ac-MTI-201 — 152 microCi intravenous solution
  Other Names: 152 microCi 225Actinium-MTI-201
  Arms: 225Ac-MTI-201 152 microCi
Drug: 254 microCi of 225Ac-MTI-201 — 254 microCi intravenous solution
  Other Names: 254 microCi 225Actinium-MTI-201
  Arms: 225Ac-MTI-201 254 microCi
Drug: 424 microCi of 225Ac-MTI-201 — 424 microCi intravenous solution
  Other Names: 424 microCi 225Actinium-MTI-201
  Arms: 225Ac-MTI-201 424 microCi
Drug: 564 microCi of 225Ac-MTI-201 — 564 microCi intravenous solution
  Other Names: 564 microCi 225Actinium-MTI-201
  Arms: 225Ac-MTI-201 564 microCi
Drug: 750 microCi of 225Ac-MTI-201 — 750 microCi intravenous solution
  Other Names: 750 microCi 225Actinium-MTI-201
  Arms: 225Ac-MTI-201 750 microCi
Drug: 998 microCi of 225Ac-MTI-201 — 998 microCi intravenous solution
  Other Names: 998 microCi 225Actinium-MTI-201
  Arms: 225Ac-MTI-201 998 microCi
Drug: 1327 microCi of 225Ac-MTI-201 — 1327 microCi intravenous solution
  Other Names: 1327 microCi 225Actinium-MTI-201
  Arms: 225Ac-MTI-201 1327 microCi

SUMMARY:
The primary aim of the study is to establish the maximum-tolerated dose (MTD) of 225Ac-MTI-201 in participants with metastatic uveal melanoma. The secondary aims are to describe the pharmacokinetics of 225Ac-MTI-201 and the toxic effects of 225Ac-MTI-201 in participants with metastatic uveal melanoma.

DETAILED DESCRIPTION:
This study will enroll patients with metastatic uveal melanoma that have failed at least one form of therapy from a single academic medical center in the United States. All participants will be informed about the study and potential risks and required to provide written informed consent prior to undergoing study-related procedures. A continual reassessment method (CRM) design will be used for this clinical trial. The study proposes single patient cohorts with dose escalation starting at 4.7 microCi of 225Ac-MTI-201 after each cohort in the absence of safety concerns (2-fold increases for doses and lower dose increases between higher doses). Dose Limiting Toxicities will be assessed using the CTCAE version 5.0 criteria.

The participants who meet the eligibility requirements will be administered a single intravenous dose of 225Ac-MTI-201. After study treatment, the study participants will stay overnight at the study center, undergo study procedures (i.e. vital signs, physical exam, multiple blood and urine sample collections) and will be scheduled to return to the clinic at 48 hours and for additional appointments weekly clinic visits the first month and on Week 9 for health status assessments, including physical exams, complete blood chemistry, and EKG. Tumor measurements every 8 weeks in first year post-injection; extended to 12 weeks in year 2; every 16 weeks in year 3, and 24 weeks in years 4 and 5. The clinic visits will involve seeing a study doctor plus radiological tests (such as MRI and/or CT scans) to see how the metastatic uveal melanoma has responded to the study drug. The protocol and informed consent documents have been reviewed and approved by the hospital human subjects review board and the study will be performed in accordance with the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic uveal melanoma.
* Progression after at least one prior line of therapy for metastatic uveal melanoma. Liver directed therapy (e.g., hepatic arterial embolization, isolated hepatic perfusion) will count as one line of therapy. Should any additional treatment(s) receive regulatory approval for metastatic uveal melanoma during the conduct of this trial, participants (if eligible for the newly approved treatment) would need to demonstrate disease progression on the additional treatment(s) before being eligible to participate in the current study. There is no limit to the number of previous treatments for metastatic disease.
* Participants must have measurable disease per RECIST 1.1.
* Adults, age 18 or over, with no upper age limit.
* ECOG (Eastern Cooperative Oncology Group) performance status of 0-1 (Karnofsky ≥ 70 percent).
* Acceptable organ and marrow function as defined below:

  * Leucocytes ≥ 3,000/μL
  * Absolute neutrophil count ≥ 1,500/μL
  * Platelets ≥ 100,000/μL
  * Aspartate aminotransferase (AST)/ Alanine aminotransferase (ALT) ≤ 2.5x institutional upper limit of normal (ULN)
  * Bilirubin ≤ 1.5x institutional upper limit of normal (ULN)
  * Creatinine clearance ≥ 60mL/min/1.73m^2 (measured by Cockcroft-Gault equation using actual body weight in kilograms, and then adjusted for body surface area)
* Male participants who are sexually active, and female participants of childbearing potential must agree to use 2 forms of FDA approved contraceptive methods during treatment with 225Ac-MTI-201 and up to 3 months following treatment.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior alpha-particle therapy.
* Has known symptomatic central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are stable without evidence of progression by imaging for at least four weeks after definitive intervention and using no more than the equivalent of dexamethasone 2 mg/d for the management of vasogenic edema, if necessary. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
* Participants with an active malignancy requiring anticancer treatment at the time of study entry that, in the judgment of the investigator could impact the results of treatment of metastatic uveal melanoma.
* Pregnant or nursing women. Women of childbearing potential (defined as having had a menstrual cycle within the past 12 months, and not having had a surgical procedure for sterilization) must have a negative pregnancy test (urine or serum) within 7 days of treatment with 225Ac-MTI-201.
* Participants with uncontrolled inter-current illness including, but not limited to, ongoing or active bacterial infection, active hepatitis B/C infection requiring antiviral therapy, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Immunocompromised participants may be at increased risk of toxicity. Therefore, HIV-positive participants, participants with acquired or congenital immunodeficiency conditions, those on chronic systemic corticosteroids requiring >10 mg of prednisone or equivalent per day will be excluded from participation. (Participants with autoimmune disease who do not require corticosteroids or are maintained on ≤10 mg of prednisone or equivalent per day ARE eligible for participation; for participants with CNS metastases on steroids, exclusion criterion bullet point #2 above will apply).
* Prior external beam radiation therapy to more than 25 percent of the bone marrow.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-07-21 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2029-02-25 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of 225Ac-MTI-201 | Within 4 weeks after study drug administration
  MTD will be determined by testing increasing doses up to 1327 microCi of 225Ac-MTI-201, administered as a single dose via IV on dose escalation cohorts 1 to 12 with 1 to 6 participants each. The MTD is reached when 6 patients receive the same highest tolerated dose of 225Ac-MTI-201. If dose-limiting toxicity (DLT) consistently occurs at the next higher dose of 225Ac-MTI-201, then 5 additional doses at the previous dose of 225Ac-MTI-201 will mark the end of clinical trial.
Number of Participants Who Experienced Dose-Limiting Toxicities (DLTs) | Within 4 weeks after study drug administration
  The following will constitute a DLT if the occurrence was within 4 weeks post-dose:
  1. Any death not due to the underlying disease or extraneous cause
  2. Absolute neutrophil count < 0.5 X 10^9/L or the development of febrile neutropenia.
  3. Grade 3 thrombocytopenia with significant bleeding, or any Grade 4 thrombocytopenia.
  4. Laboratory abnormalities that satisfy Hy's law i.e., ALT or AST elevation > 3X ULN, total bilirubin elevation > 2X ULN, absence of initial findings of cholestasis, and no other reason can be found to explain the combination of increased ALT/AST and total bilirubin
  5. Any grade 3 or higher non-hematological toxicity possibly, probably, or definitely attributed to the study drug with the following exceptions: 1) Grade 3 nausea, vomiting or diarrhea (less than 72 hours with care). 2) Grade 3 fatigue (less than 1 week). 3) Grade > 3 electrolyte abnormalities (less than 48 hours), not clinically complicated, and resolves with or without medical interventions
The Number of Participants Who Experienced Serious or Non-Serious Adverse Events | From time of signing the informed consent document until death, or lost to follow-up (approximately 3 years)
  Vital signs, physical examination, 12-lead EKG, and blood including toxicity on Days 8, 15, 22, and 29: Week 9, Follow-Up (Starting in Week 17) Adverse Event (AE), any new untoward medical occurrence or worsening of a preexisting medical condition in Participant administered study drug and that may or may not have a causal relationship with drug treatment. All AEs will be graded using the NCI CTCAE v5.0 criteria.
  Serious Adverse Event (SAE); an untoward medical occurrence at any dose that: Results in death; Is life-threatening; Requires inpatient hospitalization or causes prolongation of existing hospitalization; Results in persistent or significant disability/incapacity; Is a congenital anomaly/birth defect; Is an important medical event that may not be immediately life- threatening or result in death or hospitalization but, may jeopardize the participant or may require intervention to prevent one of the other serious outcomes; or, potential drug induced liver injury (DILI).

SECONDARY OUTCOMES:
Observed Rate of Renal Elimination of 225Ac-MTI-201 | 3 to 24 hours post-dose
  Urine samples will be obtained post-dose as needed up to 24 hours, and renal concentrations (becquerel (Bq)) over time (minutes) determined using validated method that measures 225Ac-MTI-201 radioactivity with standard Wipe Gamma Counter or a specialized gamma spectrometer. The fraction of the injected activity of the 225Ac-MTI-201 which is ultimately excreted in the urine can be then calculated.
Observed Rate of Elimination from Blood of 225Ac-MTI-201 | Prior to the initial dose on day 1; 0.042, 0.083, 0.167, 0.333, 0.667, 1.333, 2.333, 24, and 48 hours; day 8; and day 15 post-dose
  Blood samples will be obtained, and plasma concentrations (becquerel (Bq)) over time (minutes) determined using validated method that measures 225Ac-MTI-201 radioactivity with standard Wipe Gamma Counter or a specialized gamma spectrometer. The 1-compartment model will be used for describing the pharmacokinetics of 225Ac-MTI-201. The blood is set as the central compartment; elimination of 225Ac-MTI-201 from this compartment is assumed to occur through a combination of renal and hepatic elimination.
Number of Participants Who Experienced a Complete Response (CR), Partial Response (PR), Progressive Disease (PD), or Stable Disease (SD) According to Tumor Lesion Measurement | From time of signing the informed consent document until death, or lost to follow-up (approximately 3 years)
  Tumor will be measured (mm) at baseline and every 8 weeks in first year unless participant is taken off study; visit frequency is reduced in subsequent years. Follow-up visits past year-3 can be conducted via a review of clinic visit notes and/or telephone contact.
  Measurable disease is the presence of at least one measurable tumor lesion. At baseline, all lesions (up to five; maximum of two per organ) should be identified as target lesions. All other lesions (or sites of disease) including lymph nodes should be identified as non-target lesions. A lesion identified on a follow-up study not previously observed is considered a new lesion and indicates disease progression.
  CR is the loss of all target lesions. PR is at least a 30 percent decrease and PD is at least a 20 percent increase in the sum of diameters of target lesions. Stable Disease is defined as having neither sufficient shrinkage or increase to qualify for PR or PD, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Mark L McLaughlin, Study Director — Modulation Therapeutics, Inc.; Nikhil I Khushalani, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tafreshi NK, Doligalski ML, Tichacek CJ, Pandya DN, Budzevich MM, El-Haddad G, Khushalani NI, Moros EG, McLaughlin ML, Wadas TJ, Morse DL. Development of Targeted Alpha Particle Therapy for Solid Tumors. Molecules. 2019 Nov 26;24(23):4314. doi: 10.3390/molecules24234314. PMID 31779154
- [Background] Tafreshi NK, Tichacek CJ, Pandya DN, Doligalski ML, Budzevich MM, Kil H, Bhatt NB, Kock ND, Messina JL, Ruiz EE, Delva NC, Weaver A, Gibbons WR, Boulware DC, Khushalani NI, El-Haddad G, Triozzi PL, Moros EG, McLaughlin ML, Wadas TJ, Morse DL. Melanocortin 1 Receptor-Targeted alpha-Particle Therapy for Metastatic Uveal Melanoma. J Nucl Med. 2019 Aug;60(8):1124-1133. doi: 10.2967/jnumed.118.217240. Epub 2019 Feb 7. PMID 30733316
- [Background] Tafreshi NK, Kil H, Pandya DN, Tichacek CJ, Doligalski ML, Budzevich MM, Delva NC, Langsen ML, Vallas JA, Boulware DC, Engelman RW, Gage KL, Moros EG, Wadas TJ, McLaughlin ML, Morse DL. Lipophilicity Determines Routes of Uptake and Clearance, and Toxicity of an Alpha-Particle-Emitting Peptide Receptor Radiotherapy. ACS Pharmacol Transl Sci. 2021 Mar 12;4(2):953-965. doi: 10.1021/acsptsci.1c00035. eCollection 2021 Apr 9. PMID 33860213